CLINICAL TRIAL: NCT01827644
Title: A Single Center, Randomized, Open-Label, Sequential, Single Dose, 4-Period Crossover Study to Evaluate the Bioavailability and Food Effect of a Gelatin Formulation and Two Prototype Formulations of Afuresertib, an AKT Inhibitor, in Normal Healthy Volunteers
Brief Title: Bioavailability and Food Effect of the Original Gelatin Formulation and Two New Formulations of Afuresertib in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117313
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: AKT inhibitor; formulation; food effect; bioavailability; GSK2110183
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Subjects will receive single doses of AFU HPMC capsule administered in a fasted state, AFU ECT administered in a fasted state, AFU HPMC capsule administered in a fed state and AFU GC administered in a fasted state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period
  Interventions: Drug: Afuresertib GC - Fasted State; Drug: Afuresertib HPMC capsule - Fasted State; Drug: Afuresertib ECT - Fasted State; Drug: Afuresertib HPMC capsule - Fed State
- Sequence 2 (Experimental): Subjects will receive single doses of AFU ECT administered in a fasted state, AFU ECT administered in a fed state, AFU GC administered in a fasted state and AFU GC administered in a fed state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period.
  Interventions: Drug: Afuresertib GC - Fasted State; Drug: Afuresertib ECT - Fasted State; Drug: Afuresertib GC - Fed State; Drug: Afuresertib ECT - Fed State
- Sequence 3 (Experimental): Subjects will receive single doses of AFU GC administered in a fasted state, AFU GC administered in a fed state, AFU ECT administered in a fed state and AFU HPMC capsule administered in a fasted state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period.
  Interventions: Drug: Afuresertib GC - Fasted State; Drug: Afuresertib HPMC capsule - Fasted State; Drug: Afuresertib GC - Fed State; Drug: Afuresertib ECT - Fed State
- Sequence 4 (Experimental): Subjects will receive single doses of AFU GC administered in a fed state, AFU HPMC capsule administered in a fed state, AFU HPMC capsule administered in a fasted state and AFU ECT administered in a fasted state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period
  Interventions: Drug: Afuresertib HPMC capsule - Fasted State; Drug: Afuresertib ECT - Fasted State; Drug: Afuresertib GC - Fed State; Drug: Afuresertib HPMC capsule - Fed State
- Sequence 5 (Experimental): Subjects will receive single doses of AFU ECT administered in a fed state, AFU HPMC capsule administered in a fasted state, AFU GC administered in a fed state and AFU HPMC capsule administered in a fed state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period
  Interventions: Drug: Afuresertib HPMC capsule - Fasted State; Drug: Afuresertib GC - Fed State; Drug: Afuresertib HPMC capsule - Fed State; Drug: Afuresertib ECT - Fed State
- Sequence 6 (Experimental): Subjects will receive single doses of AFU HPMC capsule administered in a fed state, AFU GC administered in a fasted state, AFU ECT administered in a fasted state and AFU ECT administered in a fed state (sequentially), on Day 1 of Dosing Period 1, 2, 3 and 4 (one treatment per period) respectively, with a minimum 10 Day washout between the doses in each Dosing Period
  Interventions: Drug: Afuresertib GC - Fasted State; Drug: Afuresertib ECT - Fasted State; Drug: Afuresertib HPMC capsule - Fed State; Drug: Afuresertib ECT - Fed State

INTERVENTIONS:
Drug: Afuresertib GC - Fasted State — White opaque hard gelatin capsule containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib GC administered in fasted state
  Arms: Sequence 1; Sequence 2; Sequence 3; Sequence 6
Drug: Afuresertib HPMC capsule - Fasted State — White opaque HPMC capsule containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib HPMC capsule administered in fasted state
  Arms: Sequence 1; Sequence 3; Sequence 4; Sequence 5
Drug: Afuresertib ECT - Fasted State — White to off white, round, biconvex coated tablet containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib ECT administered in fasted state
  Arms: Sequence 1; Sequence 2; Sequence 4; Sequence 6
Drug: Afuresertib GC - Fed State — White opaque hard gelatin capsule containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib GC administered in fed state
  Arms: Sequence 2; Sequence 3; Sequence 4; Sequence 5
Drug: Afuresertib HPMC capsule - Fed State — White opaque HPMC capsule containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib HPMC capsule administered in fed state
  Arms: Sequence 1; Sequence 4; Sequence 5; Sequence 6
Drug: Afuresertib ECT - Fed State — White to off white, round, biconvex coated tablet containing afuresertib 25 mg. Subjects will receive single oral dose of afuresertib ECT administered in fed state
  Arms: Sequence 2; Sequence 3; Sequence 5; Sequence 6

SUMMARY:
This will be a randomized, open-label, sequential, single dose, 4-period crossover study. This study is being conducted to measure the relative bioavailability of the original gelatin capsule (GC) formulation and two new formulations (hydroxypropyl-methylcellulose [HPMC] capsule and enteric coated tablet [ECT]) of afuresertib (AFU), in the fed and fasted state. The study will be composed of Screening, Treatment, and Follow-up Periods. Screening assessments to determine subject eligibility will be performed within 3 weeks prior to the first dose of study drug in the Treatment Period. Eligible subjects will be randomized to receive 4 of the 6 possible study treatments (A: AFU GC administered in a fasted state, B: AFU GC administered in a fed state, C: AFU HPMC capsule administered in a fasted state, D: AFU HPMC capsule administered in a fed state, E: AFU ECT administered in a fasted state, F: AFU ECT administered in a fed state) in 4 treatment periods (one per treatment period). Subjects will receive a single dose of one of the six study treatments (A, B, C, D, E, F) on Day 1 of each Dosing Period, according to one of the 6 treatment sequences (CEDA, EFAB, ABFC, BDCE, FCBD, DAEF). There will be a minimum of 10 Day washout period between the doses administered in each Treatment Period. A Follow-up visit will be conducted within 10-14 days after the last dose. A subject's total time involved in the study will be approximately 9 weeks. At least 36 subjects will be enrolled in the study, to ensure that at least 6 subjects will be randomized to receive each treatment sequence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 40 years of age inclusive, at the time of signing the informed consent
* Body weight >=50 kilograms (kg) and body mass index (BMI) <=32 kg/m^2 (square meter)
* A female subject is eligible to participate if she is of: (A) Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea (B) Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at Screening and prior to dosing, AND: agrees to use one of the acceptable contraception methods
* Male subjects with female partners of child-bearing potential must agree to use one of the acceptable contraception methods.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QTc <450 milliseconds (msec) or QTc <480 msec in subjects with Bundle Branch Block

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of gastroesophageal reflux disease (GERD), dyspepsia, gastrointestinal (GI) bleeding, GI surgery that could affect motility
* History of atrial arrhythmias
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation
* Use of prescription or non-prescription medications, vitamins, and dietary or herbal supplements (including St John's Wort) within 7 days (or 14 days if the drug/supplement is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug until completion of the Follow-up Period, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study
* Unable to abstain from smoking tobacco or the use of nicotine-containing products while admitted to the clinic
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of Study Drug on Day 1 of Dosing Period 1, until completion of the Follow-up Period
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening
* History of heavy use of tobacco- or nicotine-containing products within 6 months prior to Screening.
* A positive drug/alcohol screen at Screening or upon check-in to the clinic on Day -1 of each Dosing Period
* A positive test for Human Immunodeficiency Virus (HIV) antibody
* Pregnant females as determined by positive serum hCG test at Screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Lactating females
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2013-07-12 (Actual); Study Completion 2013-07-12 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetics (PK) parameters of afuresertib, following administration with and without food | PK samples will be collected at Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours post-dose in each dosing period
  Relative bioavailability of afuresertib after single dose of a GC, HPMC capsule and ECT, with and without high fat/calorie meal, will be determined by the following PK parameters: Area under the plasma concentration time curve- from time zero (pre-dose) to infinite time [AUC(0-inf)] and from time zero (pre-dose) to last time of quantifiable concentration [AUC(0-t)], maximum observed plasma concentration (Cmax), time to Cmax (tmax), observed plasma concentration at 24 hours (C24), and minimal observed plasma concentration (Ct)

SECONDARY OUTCOMES:
Safety and tolerability of afuresertib as assessed by number of subjects with adverse events (AEs) | Up to 9 weeks
  AEs will be collected from the start of Study Treatment and until the Follow-up contact
Safety and tolerability of afuresertib as assessed by clinical laboratory tests | Up to 9 weeks
  Hematology, clinical chemistry and urinalysis parameters will be measured
Safety and tolerability of afuresertib as assessed by concomitant medications review | Up to 9 weeks
Safety and tolerability of afuresertib as assessed by electrocardiograms (ECG) measurements | Up to 9 weeks
  Triplicate 12-lead ECGs will be collected at Screening; on Day 1 and Day 3 of each Dosing Period; and at Follow-up
Safety and tolerability of afuresertib as assessed by vital signs measurement | Up to 9 weeks
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate
Change in phosphoAKT (pAKT) levels in peripheral blood samples following administration of a gelatin capsule, HPMC capsule and ECT | Pre-dose and 2, 12, and 24 hours post-dose in each dosing period.
  The potential relationship between plasma PK and pharmacodynamic biomarker changes (pAKT) of each formulation will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

REFERENCES:
- See also: Results for study 117313 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117313?search=study&search_terms=117313#rs